CLINICAL TRIAL: NCT06683534
Title: Use of Quercetin to Increase Resiliency to Palmitic Acid in the Human Microvasculature
Brief Title: Palmitic Acid and Human Microvascular Function
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Julie K. Freed, Executive Vice Chair, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PRO00053081
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09

CONDITIONS: Microvascular Dysfunction; Microvasculature; Cardiovascular Diseases; Cardiovascular Diseases (CVD); Microvascular Health; Obesity and Overweight
Keywords: Obesity; Supplement
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Overweight | interventions — Quercetin; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive the supplement quercetin or placebo for 30 days to determine its effect on microvascular function.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Use of oral quercetin to improve human microvascular function (Experimental): Quercetin is a non-FDA approved, over-the-counter supplement that has been shown to improve oxidative capacity in blood vessels.
  Interventions: Dietary Supplement: Quercetin (dietary supplement)
- Placebo (Placebo Comparator): A placebo will be administered for 30 days followed by assessment of the subject's microvascular function.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Quercetin (dietary supplement) — Quercetin will be provided to take one Quercetin per day for 30 days to look for differences in microvascular function.
  Arms: Use of oral quercetin to improve human microvascular function
Drug: Placebo — Subjects randomized to receive placebo will be administered a standard placebo sugar pill.
  Arms: Placebo

SUMMARY:
The goal of this study is to learn how a supplement Quercetin can affect microvascular function.

Participants will:

* give two blood draws of 5 mL each
* have a camera placed under the tongue to take pictures of blood vessels
* have 2 laser Doppler microdialysis catheters placed on the forearm to monitor blood vessels before and after local drug infusion

Researchers will compare blood vessel function of those who take estrogen supplements to those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI>30)
* Aged 18-40 years
* English Speaking

Exclusion Criteria:

* BMI>60
* Resting SBP ≥180 mmHg or DBP ≥ 110mmHg
* Pregnancy or breastfeeding.
* Prior history of myocardial infarction
* Diagnosis of more than 1 risk factor for coronary artery disease (active smoker, diabetes mellitus- type 1 or 2, congestive heart failure, hyperlipidemia, hypertension)
* Active mouth sores that affect the buccal mucosa.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood vessel dilation | 2 hours
  Peripheral microvascular dilation in response to acetylcholine, L-NAME, and sodium nitroprusside infusions will be measured using laser Doppler flowmetry with microdialysis.

SECONDARY OUTCOMES:
Change in Perfused Vessel Density | 0.5 hours
  Total vessel density (TVD) will be calculated using the DeBacker Score manual analysis on all images that have a minimum microcirculation image quality score (MIQS) of 10. Perfused vessel density (PVD) will be calculated by multiplying total vessel density (TVD) x proportion of perfused vessels (PPV%).

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Wauwatosa, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No